CLINICAL TRIAL: NCT01408394
Title: A Phase 1, Single Center, Randomized (2-Sequence), Single Blind, 3-Period Study Comparing the Safety, Tolerability, and Pharmacokinetics of Ecopipam Controlled Release Capsules With Ecopipam HCl Immediate Release Tablets in Male Adult Volunteers
Brief Title: Safety and Tolerability Comparison of Immediate and Controlled Release Formulations of Ecopipam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PSY401
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2013-05

CONDITIONS: Healthy
Keywords: safety; pharmacokinetics; controlled release; formulation
MeSH Terms: interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg immediate release form (Active Comparator): This is the formulation currently in use
  Interventions: Drug: Ecopipam immediate release form
- 90 mg controlled release (Experimental): This is the low dose of the controlled release form
  Interventions: Drug: 90 mg controlled release form
- 180 mg controlled release form (Experimental): This is the medium controlled release dose
  Interventions: Drug: 180 mg controlled release form

INTERVENTIONS:
Drug: Ecopipam immediate release form — Tablet containing 100 mg of the immediate release form of ecopipam
  Other Names: SCH 39166; PSYRX101
  Arms: 100 mg immediate release form
Drug: 90 mg controlled release form — This is the 90 mg controlled release form
  Other Names: SCH 39166; PSYRX101
  Arms: 90 mg controlled release
Drug: 180 mg controlled release form — This is the 180 mg controlled release capsule
  Other Names: SCH 39166; PSYRX101
  Arms: 180 mg controlled release form

SUMMARY:
Ecopipam hydrochloride (HCl) is an investigational drug being studied for several possible diseases. To date, all clinical studies have been done using the ecopipam immediate release (IR) tablet. However, a controlled release (CR) capsule formulation of ecopipam has been produced that may be able to improve its effectiveness and reduce its side effects. The main purpose of this study is to evaluate the safety and tolerability of ecopipam CR capsules when given as single oral dose in healthy volunteers.

DETAILED DESCRIPTION:
Ecopipam hydrochloride (HCl) is an investigational drug being studied for several possible diseases. To date, all clinical studies have been done using the ecopipam immediate release (IR) tablet. However, a controlled release (CR) capsule formulation of ecopipam has been produced that may be able to improve its effectiveness and reduce its side effects. The main purpose of this study is to evaluate the safety and tolerability of ecopipam CR capsules when given as single oral dose in healthy volunteers. Another purpose of the study is to measure how much CR and IR ecopipam gets into the blood stream, and how long the body takes to get rid of them. Information about any side effects that may occur will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated, IRB-approved informed consent form before any protocol-specific screening procedures
2. Non-smoking male subjects between the ages of 18 and 45 years (inclusive)
3. In good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation
4. Willing and able to complete all study assessments and procedures
5. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and a weight between 65 and 100 kg (inclusive)
6. QTcB interval (Bazett's correction factor) of the baseline ECG must be ≤ 450 ms at screening

Exclusion Criteria:

1. Subjects with a history of suicide attempt or with past or current active suicidal ideation
2. Subjects with a history of seizures or with head trauma leading to loss of consciousness
3. Subjects with clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
4. History of any primary malignancy, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years
5. Supine blood pressure >140/90 mm/Hg or resting heart rate ≥100 bpm at the screening visit
6. History of substance-related disorders (with the exception of caffeine-related and nicotine-related disorders) or eating disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) within 1 year of screening
7. History of smoking or the use of nicotine containing products within 3 months of screening by self reporting
8. A positive alcohol Breathalyzer or urine drug screen for drugs of abuse at the screening visit or at the beginning of the inpatient period
9. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of the screening period
10. Treatment with any other prescription or non-prescription drugs (including vitamins, herbal, and dietary supplements) within 7 days or 5 half-lives of the screening visit, whichever is longer. Acetaminophen will be permitted for intermittent treatment at doses of less than 2 grams/day
11. Subjects with a history of previous administration of ecopipam or of an allergic reaction or hypersensitivity to any drug or to any component of the CR formulation
12. Blood collection or blood loss of greater than 500 mL within 56 days prior to screening
13. Positive for human immunodeficiency virus (HIV) at screening
14. Positive for Hepatitis B surface antigen (HbsAg) or positive Hepatitis C virus (HCV) antibody at screening
15. Any other condition and/or situation that causes the investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety | 0-48 hours
  Physical examinations, adverse events, vital signs, clinical laboratory values, ECG and Columbia Suicide Severity Ratings scale

SECONDARY OUTCOMES:
Pharmacokinetics | 0-48 hours
  Pharmacokinetic properties of CR and IR ecopipam following oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MB,ChB,FACP, Principal Investigator — SNBL Clinical Pharmacology Center, Inc.
Locations (1):
- SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States